## Moderation analysis of the MI-NAV trial: statistical analysis plan

Clinical trials registration number: NCT03871712
SAP version: 1st version
Date: 17.05.2023

This document is a statistical analysis plan for a moderation analysis of the MI-NAV trial. Detailed information on the MI-NAV trial, including primary analyses can be found in the trial article:

Aanesen F, Grotle M, Rysstad TL, et al. Effectiveness of adding motivational interviewing or a stratified vocational advice intervention to usual case management on return to work for people with musculoskeletal disorders: the MI-NAV randomised controlled trial. *Occupational and Environmental Medicine* 2023;**80**:42-50.

#### **Contributors:**

Martjie Venter,<sup>1</sup> Margreth Grotle,<sup>2,3</sup> Britt Elin Øiestad,<sup>4</sup> Fiona Aanesen,<sup>5</sup> Alexander Tingulstad,<sup>4</sup> Tarjei Rysstad,<sup>4</sup> Michael Ferraro,<sup>1,6</sup> James H McAuley,<sup>1,6</sup> Aidan G Cashin<sup>1,6</sup>

<sup>&</sup>lt;sup>1</sup>Centre for Pain IMPACT, Neuroscience Research Australia, Australia

<sup>&</sup>lt;sup>2</sup> Centre for Intelligent Musculoskeletal Health, Department of Rehabilitation Science and Health Technology, Oslo Metropolitan University, Oslo, Norway

<sup>&</sup>lt;sup>3</sup> Research and Communication Unit for MSK Health (FORMI), Division of Clinical Neuroscience, Oslo University Hospital, Oslo, Norway

<sup>&</sup>lt;sup>4</sup> Department of Rehabilitation Science and Health Technology, Oslo Metropolitan University, Oslo, Norway

<sup>&</sup>lt;sup>5</sup> National Institute of Occupational Health, Oslo, Norway

<sup>&</sup>lt;sup>6</sup> School of Health Sciences, University of New South Wales, Australia

The MI-NAV trial (1) was a three-arm parallel pragmatic randomised controlled trial evaluating the effectiveness of two vocational treatment packages (MI, motivational interviewing plus usual case management; SVAI, stratified vocational advice intervention plus usual case management) compared to usual case management alone, on sickness absence days among 514 people on sick leave due to musculoskeletal disorders. The MI-NAV trial showed that adding MI or a SVAI to usual case management resulted in a non-statistically significant reduction in seven sickness absence days over 6 months for workers on sick leave due to musculoskeletal disorders in Norway. The trial findings were uncertain due to wide confidence intervals. To determine if potential relationship between the intervention and the outcome depends on the value of a third factor, moderation analysis can be conducted. This information can be used to tailor treatments to specific patient populations, leading to better clinical outcomes. Therefore, this statistical analysis plan describes the planned moderation analysis of the MI-NAV trial.

## **Primary objective**

The primary objective in this study is to assess any moderation of the two vocational treatment effects by considering a set of plausible baseline patient characteristics. We aim to identify the characteristics of sick listed workers due to musculoskeletal disorders who are more likely to benefit from either MI or SVAI.

## **Primary outcome**

The primary outcome for the MI-NAV trial and for this study is sickness absence days, measured as the number of sickness absence days from baseline assessment date until the six-month follow-up. Sickness absence days will be calculated from information provided by different national registries including information on sick leave payments, sick leave certificates, work assessment allowance, disability pensions and employment percentage. To convert time on sick leave to actual time away from work we will account for the participants' contracted work hours and the amount of sick leave. This will be summed up and converted to sickness absence days, according to a 5-day working week when working full-time.

# Moderators

Potential treatment effect modifiers for this study are presented in Table 1. The selection of potential treatment effect modifiers for this study was based on published literature investigating treatment moderators in musculoskeletal disorders, prognostic cohort studies, and theoretical support.

**Table 1.** Potential treatment effect modifiers

| Variable | Description/ categories | Evidence to support | Hypothesis direction |
|---|---|---|---|
| Age (18-67 years) | Continuous, years | Gurung et al.,2015 (2) | Younger > Older |
| | | Garcia et al., 2016 (3) | |
| | | Broderick et al., 2016 (4) | |
| Gender | Male | Gurung et al.,2015 (2) | Female > Male |
| | Female | | |
| | | Hee et al,. 2021 (5) | |
| Education | Lower Education | Gurung et al.,2015 (2) | Higher level of education > Lower level of |
| | Higher Education | | education |
| | | Broderick et al., 2016 (4) | |
| | | Roseen et al., 2021 (6) | |
| | | Beneciuk et al., 2017 (7) | |
| Smoking Status | Non-smoker | Roseen et al., 2021 (6) | Non-smoker > Smoker |
| | Smoker | | |
| | | Beneciuk et al., 2023 (8) | |
| | | D- 7tt -1 2024 (0) | |
| | 0 1 | De Zoete et al., 2021 (9) | AL LONGLAN LONGLAN |
| Body Mass Index (BMI) | Continuous, number | Hayden et al., 2020 (10) | Normal BMI > Abnormal BMI |
| Type of Work | White collar<br>Blue Collar | Gurung et al.,2015 (2) | White collar > Blue collar |
| | Blue Collar | | |
| | | Hayden et al., 2020 (10) | |
| Distress | Continuous, 0-10 scale | Gurung et al.,2015 (2) | Low distress > Increased distress |
| ((1) | (higher scores indicate | | |
| "How much have you | more distress) | Hee et al,. 2021 (5) | |
| been bothered by | | | |
| feeling depressed in the past week?" | | | |
| pasi week? | | | |

| Continuous, 0-10 scale | Gurung et al.,2015 (2) | Lower Pain intensity > Pain intensity |
|---|---|---|
| , , | | |
| worse pain) | Hahne et al., 2017 (11) | |
| | Kuijer et al., 2006 (12) | |
| | Jensen et al., 2013 (13) | |
| Continuous, 0-10 scale | | |
| - | , , , , | |
| better return to work | Kuijer et al., 2006 (12) | |
| expectancy) | | |
| | Jensen et al., 2013 (13) | |
| Yes | Gurung et al.,2015 (2) | No medication > Medication use |
| No | | |
| | Roseen et al., 2021 (6) | |
| | Beneciuk et al., 2017 (7) | |
| | Beneciuk et al., 2023 (8) | |
| | Hayden et al., 2020 (10) | |
| Norwegian<br>Other | Campbell & Edwards., 2012 (15) | Norwegian > Other |
| | Fillingim, 2016 (16) | |
| Continuous, days | Dekkers- Sánchez et al., 2008 (17) | Less previous sickness absence > Increased previous sickness absence |
| Continuous, 0-100 scale | Laaksonen et al., 2011(18) | Greater self-perceived health > Reduced |
| (higher scores indicate | | self-perceived health. |
| better perceived health) | | |
| | (higher scores indicate worse pain) Continuous, 0-10 scale (higher scores indicate better return to work expectancy) Yes No Norwegian Other Continuous, days Continuous, 0-100 scale (higher scores indicate | (higher scores indicate worse pain) Hahne et al., 2017 (11) Kuijer et al., 2006 (12) Jensen et al., 2013 (13) Continuous, 0-10 scale (higher scores indicate better return to work expectancy) Jensen et al., 2006 (12) Kuijer et al., 2006 (14) Kuijer et al., 2006 (14) Kuijer et al., 2006 (12) Kuijer et al., 2006 (12) Sensen et al., 2013 (13) Yes No Roseen et al., 2013 (13) Yes No Roseen et al., 2021 (6) Beneciuk et al., 2021 (6) Beneciuk et al., 2023 (8) Hayden et al., 2020 (10) Norwegian Other Fillingim, 2016 (16) Continuous, days Continuous, 0-100 scale (higher scores indicate Laaksonen et al., 2011(18) |

## Statistical analysis

Baseline demographic and clinical characteristics will be summarized using counts and percentages for categorical variables and means and standard deviations or median and interquartile range for continuous variables.

We will investigate any potential modification of the effect of MI vs UC and SVAI vs UC separately considering the set of plausible patient characteristics. To identify potential effect modifiers, we will conduct a formal moderation analysis using a test for statistical interaction (19, 20). We will create separate linear regression models for each potential moderator variable for each intervention comparison investigating *treatment modification* by incorporating a group x potential moderator interaction term. Specifically, we will build each model including a term for the outcome sickness absence days, group allocation, potential modifier, and a group allocation x potential modifier interaction term. We will estimate the treatment effect, 95% confidence interval and p-value for each potential modifier interaction. Interaction coefficients for dichotomous variables will be interpreted as the effect of the vocational intervention, relative to usual case management comparison, in those with the baseline characteristic compared with those who do not have the characteristic. Interaction coefficients for continuous variables will be interpreted as the additional benefit of the vocational intervention, relative to the usual case management comparison, for every one-unit increase in the continuous variable. All statistical analyses will be conducted using R.

#### Missing data

We will assess the proportion and patterns of missing moderator and outcome data. We will conduct all analyses on complete cases if the proportion of missing data is less than 5% for any of the moderators or outcome. If missing data exceeds 5%, we will use multiple imputations by chain equations to impute datasets using the 'mice' package.

#### References

- 1. Aanesen F, Grotle M, Rysstad TL, Tveter AT, Tingulstad A, Løchting I, et al. Effectiveness of adding motivational interviewing or a stratified vocational advice intervention to usual case management on return to work for people with musculoskeletal disorders: the MI-NAV randomised controlled trial. Occup Environ Med. 2023;80(1):42-50.
- 2. Gurung T, Ellard DR, Mistry D, Patel S, Underwood M. Identifying potential moderators for response to treatment in low back pain: A systematic review. Physiotherapy. 2015;101(3):243-51.
- 3. Garcia AN, Costa Lda C, Hancock M, Costa LO. Identifying Patients With Chronic Low Back Pain Who Respond Best to Mechanical Diagnosis and Therapy: Secondary Analysis of a Randomized Controlled Trial. Phys Ther. 2016;96(5):623-30.
- 4. Broderick JE, Keefe FJ, Schneider S, Junghaenel DU, Bruckenthal P, Schwartz JE, et al. Cognitive behavioral therapy for chronic pain is effective, but for whom? Pain. 2016;157(9):2115-23.
- 5. Hee SW, Mistry D, Friede T, Lamb SE, Stallard N, Underwood M, et al. Identification of subgroup effect with an individual participant data meta-analysis of randomised controlled trials of three different types of therapist-delivered care in low back pain. BMC Musculoskelet Disord. 2021;22(1):191.
- 6. Roseen EJ, Gerlovin H, Felson DT, Delitto A, Sherman KJ, Saper RB. Which Chronic Low Back Pain Patients Respond Favorably to Yoga, Physical Therapy, and a Self-care Book? Responder Analyses from a Randomized Controlled Trial. Pain Med. 2021;22(1):165-80.
- 7. Beneciuk JM, Hill JC, Campbell P, Afolabi E, George SZ, Dunn KM, et al. Identifying Treatment Effect Modifiers in the STarT Back Trial: A Secondary Analysis. J Pain. 2017;18(1):54-65.
- 8. Beneciuk JM, George SZ, Patterson CG, Smith CN, Brennan GP, Wegener ST, et al. Treatment effect modifiers for individuals with acute low back pain: secondary analysis of the TARGET trial. Pain. 2023;164(1):171-9.
- 9. de Zoete A, de Boer MR, Rubinstein SM, van Tulder MW, Underwood M, Hayden JA, et al. Moderators of the Effect of Spinal Manipulative Therapy on Pain Relief and Function in Patients with Chronic Low Back Pain: An Individual Participant Data Meta-analysis. Spine (Phila Pa 1976). 2021;46(8):E505-e17.
- 10. Hayden JA, Wilson MN, Stewart S, Cartwright JL, Smith AO, Riley RD, et al. Exercise treatment effect modifiers in persistent low back pain: an individual participant data meta-analysis of 3514 participants from 27 randomised controlled trials. Br J Sports Med. 2020;54(21):1277-8.
- 11. Hahne AJ, Ford JJ, Richards MC, Surkitt LD, Chan AYP, Slater SL, et al. Who Benefits Most From Individualized Physiotherapy or Advice for Low Back Disorders? A Preplanned Effect Modifier Analysis of a Randomized Controlled Trial. Spine (Phila Pa 1976). 2017;42(21):E1215-e24.
- 12. Kuijer W, Groothoff JW, Brouwer S, Geertzen JH, Dijkstra PU. Prediction of sickness absence in patients with chronic low back pain: a systematic review. J Occup Rehabil. 2006;16(3):439-67.
- 13. Jensen OK, Stengaard-Pedersen K, Jensen C, Nielsen CV. Prediction model for unsuccessful return to work after hospital-based intervention in low back pain patients. BMC Musculoskeletal Disorders. 2013;14(1):140.
- 14. Hagen E, Svensen E, Eriksen H. Predictors and Modifiers of Treatment Effect Influencing Sick Leave in Subacute Low Back Pain Patients. Spine. 2006;30:2717-23.

- 15. Campbell CM, Edwards RR. Ethnic differences in pain and pain management. Pain Manag. 2012;2(3):219-30.
- 16. Fillingim RB. Individual differences in pain: understanding the mosaic that makes pain personal. Pain. 2017;158 Suppl 1(Suppl 1):S11-s8.
- 17. Dekkers-Sánchez PM, Hoving JL, Sluiter JK, Frings-Dresen MHW. Factors associated with long-term sick leave in sick-listed employees: a systematic review. Occupational and Environmental Medicine. 2008;65(3):153.
- 18. Laaksonen M, Kääriä SM, Leino-Arjas P, Lahelma E. Different domains of health functioning as predictors of sickness absence--a prospective cohort study. Scand J Work Environ Health. 2011;37(3):213-8.
- 19. Pincus T, Miles C, Froud R, Underwood M, Carnes D, Taylor SJ. Methodological criteria for the assessment of moderators in systematic reviews of randomised controlled trials: a consensus study. BMC Med Res Methodol. 2011;11:14.
- 20. Sun X, Briel M, Walter SD, Guyatt GH. Is a subgroup effect believable? Updating criteria to evaluate the credibility of subgroup analyses. Bmj. 2010;340:c117.